CLINICAL TRIAL: NCT01193140
Title: An Extension Study to Evaluate the Safety of Veliparib in Combination With Temozolomide in Subjects With Solid Tumors.
Brief Title: To Evaluate the Safety of Veliparib in Combination With Temozolomide in Subjects With Solid Tumors
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Abbott (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: M12-273
Record Dates: First submitted 2010-07-28; First posted 2010-09-01 (Estimated); Last update posted 2012-11-21 (Estimated); Status verified 2012-11

CONDITIONS: Solid Tumor Cancers
Keywords: veliparib; relapsed and refractory tumors; Temodar; temozolomide; ABT-888; Solid Tumors
MeSH Terms: conditions — Recurrence; Neoplasms | interventions — veliparib; Temozolomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Arm A (Experimental)
  Interventions: Drug: veliparib; Drug: Temozolomide

INTERVENTIONS:
Drug: veliparib — Dose orally twice daily for 7 days, consecutively, every cycle
  Other Names: ABT-888
Drug: Temozolomide — Dose orally once daily for 5 days, consecutively, every cycle
  Other Names: Temodar

SUMMARY:
To evaluate the safety and tolerability of the veliparib/TMZ combination in subjects with solid tumors.

DETAILED DESCRIPTION:
An extension study to evaluate the safety of veliparib in combination with temozolomide in subjects with solid tumors

ELIGIBILITY:
Inclusion Criteria

1. Subject has completed study participation in Study M11-846
2. Eastern Cooperative Oncology Group (ECOG) performance score of 0 to 2.
3. Subject must have adequate hematologic, renal and hepatic function per institutional normal range as follows: • Bone Marrow: Absolute neutrophil count (ANC ≥ 1,500/mm3 (1.5 × 109/L); Platelets ≥ 100,000/mm3 (100 × 109/L); Hemoglobin ≥ 9.5 g/dL (1.4 mmol/L); • Renal function: Serum creatinine ≤ 1.5 × upper limit of normal (ULN) range OR creatinine clearance ≥ 50 mL/min/1.73 m2 for subjects with creatinine levels above institutional normal; • Hepatic function: AST and ALT ≤ 2.5 × the ULN range. For subjects with liver metastases, AST and ALT < 5 × the ULN range; Bilirubin ≤ 1.5 × the ULN range. • Partial Thromboplastin Time (PTT) must be ≤ 1.5 × the ULN range and INR < 1.5. Subjects on anticoagulant therapy (such as Coumadin) will have an appropriate PTT and INR as determined by the Investigator.
4. Women of childbearing potential must agree to use adequate contraception (one of the following listed below) prior to study entry, for the duration of study participation and for 90 days following completion of therapy. Women of childbearing potential must have a negative serum pregnancy test within 28 days prior to initiation of treatment and a negative urine pregnancy test on Cycle 1 Day 1 and/or post menopausal women must be amenorrheic for at least 12 months to be considered of non-childbearing potential. • Total abstinence from sexual intercourse (minimum one complete menstrual cycle); • Vasectomized partner; • Hormonal contraceptives (oral, parenteral or transdermal) for at least 3 months prior to study drug administration; • Double-barrier method (condoms, contraceptive sponge, diaphragm or vaginal ring with spermicidal jellies or cream); • IUD (Intrauterine Device).

Exclusion Criteria

1. Subject has received anticancer agent(s) or an investigational agent (except for veliparib) within 28 days prior to study drug administration. Subjects who have not recovered to within one grade level (not to exceed grade 2) of their baseline following a significant adverse event or toxicity attributed to previous anticancer treatment are excluded.
2. Subject has undergone major surgery within the previous 28 days prior to study drug administration.
3. Subject has received radiotherapy within 28 days prior to study drug administration.
4. Clinically significant and uncontrolled major medical condition(s) including but not limited to: • Active uncontrolled infection; • Symptomatic congestive heart failure;• Unstable angina pectoris or cardiac arrhythmia; • Psychiatric illness/social situation that would limit compliance with study requirements; • Any medical condition, which in the opinion of the Study Investigator, places the subject at an unacceptably high risk for toxicities.
5. Subject is pregnant or lactating.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2010-07; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
To evaluate the safety and tolerability of veliparib/TMZ combination in subjects with solid tumors | Continuous starting with Day1 and 30 Days following last dose.
  Safety and tolerability will be assessed through clinical laboratory tests, electrocardiograms (ECGs), vital signs, physical exams and adverse event assessments

SECONDARY OUTCOMES:
To assess effect of veliparib/TMZ combination regimen on progression free survival, overall survival, the objective response rate, time to progression and Eastern Cooperative Oncology Group (ECOG) performance status in subjects with solid tumors | Every 12 weeks from Day1 and continuing up to 18 months following last dose.

CONTACTS AND LOCATIONS:
Overall Officials: Bhardwaj Dessai, MD, Study Director — Abbott
Locations (2):
- United States (2):
  - Site Reference ID/Investigator# 43022, Encinitas, California
  - Site Reference ID/Investigator# 42662, Santa Monica, California